CLINICAL TRIAL: NCT05401630
Title: Mental Stress Reactivity in Women With Coronary Microvascular Dysfunction
Brief Title: Mental Stress Reactivity in Women With CMD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Puja Mehta, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY00003154; 1R01HL157311-01A1 (NIH); 2025P012678 (Other: Emory IRB)
Record Dates: First submitted 2022-05-10; First posted 2022-06-02 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Post-menopause
Keywords: Microvascular; Sympathetic activity; Mental Stress; Angina
MeSH Terms: conditions — Stress, Psychological; Angina Pectoris | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Symptomatic women with no obstructive CAD who have CMD (Experimental): Symptomatic women with chest pain and no obstructive CAD who have an abnormal myocardial flow reserve (MFR < 2.5)
  Interventions: Other: Study Procedures
- Symptomatic women with chronic obstructive CAD (oCAD) (Experimental): This group will serve as one comparison group since these women represent the prevailing paradigm of ischemia from obstructive stenosis while sharing common cardiovascular risk factors with the CMD group.
  Interventions: Other: Study Procedures
- Asymptomatic control women with no prior history of CAD or angina (Active Comparator): Asymptomatic control women with no prior history of CAD or angina, who are age-matched to the CMD women; not on any cardiac medications, who will also have to pass a maximal Bruce protocol exercise treadmill test.
  Interventions: Other: Study Procedures

INTERVENTIONS:
Other: Study Procedures — All participants will answer a series of questionnaires that address several factors such as patient medical history, family history, medication usage, health behaviors, psychological factors, etc. Questionnaires related to symptoms, psychological factors, depression, anxiety, and quality of life will be taken.
  All participants will undergo 123I-MIBG SPECT imaging in the morning in a fasting state. Mental Stress Testing will be conducted in the Laboratory in the morning after fasting for at least 4 hours and withdrawal of all vasoactive medications, caffeine, and tobacco 24-48 hours before testing. Participants will also undergo 1-week of Home Monitoring using a single-use, noninvasive, water-resistant, 7-day ambulatory ECG monitoring, which offers the advantage of direct access to raw data that can be downloaded from the device after use.
  A 3-day food recall diary, cognitive assessments via the NIH Toolbox, and a Sleep diary during home monitoring will be collected.

SUMMARY:
Coronary Microvascular Dysfunction (CMD) occurs when there are problems in the small blood vessels/arteries of the heart, resulting in persistent chest pain that affects women.

There are an estimated 3 million women in the US with CMD and about 100,000 new cases annually. This research will investigate whether the stress response physiology and autonomic function in response to mental stress are different in women with CMD compared to other groups. The autonomic nervous system (ANS) controls normally involuntary activities, such as heart rate, respiration (breathing), body temperature, blood pressure, and urinary function. This study will also examine how chronic and daily life mental stress affects the heart and blood vessels.

Participants from this study will be recruited mainly from Emory Healthcare-associated hospitals, the Emory Heart Disease Center for Prevention, and Emory Healthcare outpatient cardiology clinics. Participants will have physical exams, blood tests, stress tests, exercise tests, surveys, questionnaires, and images taken of their hearts and blood vessels. They will be asked to take home devices to monitor their autonomic function, sleep, and track their mood, stress level, and symptoms for one week. Data and specimens will be saved for future research.

DETAILED DESCRIPTION:
The overall goal of this project is to clarify the mechanisms and pathophysiology of how psychological stress contributes to Major Adverse Cardiovascular Events (MACE) in women despite having no obstructive CAD. Through this proposal, the research team expects to have an improved understanding of the relationships between mental stress and coronary microvascular dysfunction in women.

One-third to one-half of women with chest pain who are suspected of having myocardial ischemia and undergo coronary angiography are actually found to have no obstructive coronary artery disease (CAD) (<50% luminal stenosis) and thus are often reassured and dismissed without a cardiac diagnosis or therapy. Current evidence suggests that a large proportion of these women have coronary microvascular dysfunction (CMD) and are at significantly increased risk of major adverse cardiovascular events (MACE), including myocardial infarction, heart failure, and sudden cardiac death. However, because of substantial knowledge gaps, these patients also have recurrent hospitalizations for chest pain, reduced health-related quality of life, and comparable disability and healthcare costs to obstructive CAD patients. Cardiac rest/stress positron emission tomography (PET) imaging can detect impaired myocardial flow reserve (MFR) and diagnose CMD. However, therapeutic strategies are poorly developed, with limited studies to inform clinicians on the treatment of CMD.

Comorbid psychological factors such as anxiety and depression are prevalent in women with persistent angina, and stress can contribute to and exacerbate angina, implicating the autonomic nervous system (ANS) as one mechanistic pathway in CMD-related ischemia and MACE. The preliminary data indicate that women with CMD have ANS dysfunction with sympathetic predominance compared to non-CMD controls. The research team has shown that women have more mental stress ischemia (MSI) and stress-induced peripheral microvascular vasoconstriction compared to men. MSI is an important prognostic marker with an estimated two-fold increase in MACE, including mortality, regardless of the severity of CAD.

The research team posits that an improved understanding of psychological stress reactivity in CMD patients will help tease out the underlying mechanisms contributing to adverse outcomes in CMD-related ischemia and provide new treatment targets to reduce symptom burden and MACE. The overall goal of this project is to clarify the mechanisms and pathophysiology of how psychological stress contributes to MACE in women despite having no obstructive CAD. The research team has also shown that coronary microvascular responses to mental stress are reflected in the peripheral microvascular circulation. This proposal addresses an important knowledge gap in an understudied population and is a direct extension of their prior work. Findings from this work have the potential to inform therapeutic strategies in CMD, a problem that impacts an estimated 3 million American women. The unifying hypothesis is that women with CMD have exaggerated sympathetic activation and abnormal vasoreactivity to mental stress, which predisposes them to adverse outcomes even in the absence of obstructive CAD.

Three groups of post-menopausal women will be compared: (1) symptomatic women with no obstructive CAD who have CMD ; (2) symptomatic women with chronic obstructive CAD (oCAD); and (3) asymptomatic control women with no prior history of CAD or angina, who are age-matched to the CMD women. The oCAD group will serve as a comparison group since these women represent the prevailing paradigm of ischemia from obstructive stenosis while sharing common cardiovascular risk factors that could confound the findings.

No study has comprehensively characterized mental stress reactivity by pairing autonomic responses and vascular reactivity in women with CMD, and with follow-up of angina and quality of life (QoL). This study would provide critical data on the clinical significance of these measures in the CMD population.

ELIGIBILITY:
CMD Group

Inclusion Criteria:

* Symptomatic postmenopausal women with chest pain
* age≥45 years old
* willing to undergo cardiac MIBG scan
* willing to undergo mental stress testing
* competent to give informed consent

Exclusion Criteria:

* Significant epicardial stenosis (defined by coronary stenosis ≥ 70% in any epicardial coronary artery or hemodynamically significant stenosis determined by fractional flow reserve)
* Left ventricular systolic dysfunction (ejection fraction ≤ 50%)
* Heart failure with a preserved ejection fraction
* Significant anemia or blood dyscrasia
* Severe uncontrolled hypertension >180/100
* Unable to lie flat for mental stress testing
* Pre-menopausal
* Pregnant
* Pericarditis/myocarditis
* History of percutaneous coronary intervention
* Coronary artery bypass grafting
* Acute myocardial infarction/acute coronary syndrome/unstable angina within 1 month
* Significant valvular disease, including aortic or mitral stenosis
* Sinus node dysfunction/pacemaker, 2nd or 3rd-degree atrioventricular block
* Severe lung, renal, liver, or psychiatric illness
* Current neoplasm
* History of substance abuse
* Acute illness such as infection in the previous 4 weeks
* Life-expectancy less than 2 years
* Unable to safely withdraw medications for mental stress testing
* Significant psychiatric illness that precludes safe participation in the study
* Conditions that preclude accurate or safe testing and patient refusal
* Unable to consent

Obstructive CAD (oCAD) Group

Inclusion Criteria:

* Symptomatic postmenopausal women with chest pain who have obstructive CAD in at least one epicardial coronary artery
* willing to undergo cardiac MIBG scan
* willing to undergo mental stress testing
* competent to give informed consent

Exclusion Criteria:

* Significant epicardial stenosis (defined by coronary stenosis ≥ 70% in any epicardial coronary artery or hemodynamically significant stenosis determined by fractional flow reserve)
* Left ventricular systolic dysfunction (ejection fraction ≤ 50%)
* Heart failure with a preserved ejection fraction
* Significant anemia or blood dyscrasia
* Severe uncontrolled hypertension >180/100
* Unable to lie flat for mental stress testing
* Pre-menopausal
* Pregnant
* Pericarditis/myocarditis
* History of percutaneous coronary intervention
* Coronary artery bypass grafting
* Acute myocardial infarction/acute coronary syndrome/unstable angina within 1 month
* Significant valvular disease, including aortic or mitral stenosis
* Sinus node dysfunction/pacemaker, 2nd or 3rd-degree atrioventricular block
* Severe lung, renal, liver, or psychiatric illness
* Current neoplasm
* History of substance abuse
* Acute illness such as infection in the previous 4 weeks
* Life expectancy is less than 2 years
* Unable to safely withdraw medications for mental stress testing
* Significant psychiatric illness that precludes safe participation in the study
* Conditions that preclude accurate or safe testing and patient refusal
* Unable to consent

Asymptomatic Control Group

Inclusion Criteria:

* Asymptomatic postmenopausal women, age ≥ 45 years old
* Healthy volunteer with no cardiac risk factors
* No history or diagnosis of heart disease
* Not on any cardiac medications
* Normal maximal exercise treadmill stress testing (ETT)
* Fully understanding and willing to undergo mental stress testing
* Willing to sign the informed consent

Exclusion Criteria:

* Significant epicardial stenosis (defined by coronary stenosis ≥ 70% in any epicardial coronary artery or hemodynamically significant stenosis determined by fractional flow reserve)
* Left ventricular systolic dysfunction (ejection fraction ≤ 50%)
* Heart failure with a preserved ejection fraction
* Significant anemia or blood dyscrasia
* Severe uncontrolled hypertension >180/100
* Unable to lie flat for mental stress testing
* Pre-menopausal
* Pregnant
* Pericarditis/myocarditis
* History of percutaneous coronary intervention
* Coronary artery bypass grafting
* Acute myocardial infarction/acute coronary syndrome/unstable angina within 1 month
* Significant valvular disease, including aortic or mitral stenosis
* Sinus node dysfunction/pacemaker, 2nd or 3rd-degree atrioventricular block
* Severe lung, renal, liver, or psychiatric illness
* Current neoplasm
* History of substance abuse
* Acute illness such as infection in the previous 4 weeks
* Life expectancy is less than 2 years
* Unable to safely withdraw medications for mental stress testing
* Significant psychiatric illness that precludes safe participation in the study
* Orthopedic limitation that will prevent ETT
* LDL >120 mg/dL
* Fasting blood glucose >95 mg/dL
* Hypertension, defined as resting BP >120/80
* Diabetes
* Hyperlipidemia
* Smoking
* Conditions that preclude accurate or safe testing and patient refusal
* Unable to consent

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 150 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Planar late Heart to Mediastinal Ratio (MIBG imaging) | At the end of MIBG procedure
  The research team will compare resting sympathetic activity measured with 123I-meta-iodobenzylguanidine (MIBG) imaging between CMD women and the two control groups. The heart to the mediastinal ratio (HMR) which is an index of MIBG uptake will be calculated as per standard methods. The HMR reflects norepinephrine kinetics. Higher sympathetic activity and turnover cause less MIBG to be retained and result in a lower HMR. MIBG SPECT defect score will be determined by late (4 hours) MIBG uptake by visual blind scoring using the standard 17-segment model with 0=normal tracer uptake, 1=mildly reduced uptake, 2=moderately reduced uptake, 3=severely reduced uptake, 4=absent tracer uptake, as defined by Bax et al.
Changes in HRV with mental stress | Baseline (prior to stress testing) and during mental stress test
  The research team will also compare autonomic reactivity during a standardized mental stress test, including heart rate variability (HRV) between CMD women and the two control groups
Changes in pre-ejection period (PEP) with mental stress | Baseline (prior to stress testing) and during mental stress test
  The research team will also compare autonomic reactivity during a standardized mental stress test, including the pre-ejection period (PEP) between CMD women and the two control groups. This measures systolic time interval and reflects cardiac contractility (which is under the beta-adrenergic influence). Impedance ECG measures PEP from the onset of ventricular depolarization (Q-wave on ECG) to the opening of the aortic valve for ejection of blood from the left ventricle.

SECONDARY OUTCOMES:
Changes in flow mediated dilation (FMD test) to acute mental stress in CMD women. | Baseline (prior to stress testing) and at the end of the mental stress test
  The research team will compare peripheral microvascular vasoconstriction during mental stress, as well as changes in peripheral microvascular function and flow-mediated dilation with mental stress, between CMD women and the two control groups. Readings of blood flow in one of the arteries of the arm using an ultrasound. Then a blood pressure cuff will be placed around the forearm and will be inflated to stop the flow of blood for 5 minutes. After 5 minutes, the blood pressure cuff will be deflated and the readings taken again.
Changes in Peripheral arterial tonometry (PAT) test to acute mental stress in CMD women. | Baseline (prior to stress testing) and at the end of the mental stress test
  The research team will compare peripheral microvascular vasoconstriction during mental stress, as well as changes in peripheral microvascular function and flow-mediated dilation with mental stress, between CMD women and the two control groups. A blood pressure cuff will be placed on one arm, and probes will be placed on the fingers. In order to get a good tracing, the participant will need to remain quiet and very still for at least 5 minutes. Then, the blood pressure cuff will be inflated for 5 minutes, and more recordings will be done. At the end of the 5 minutes, the blood pressure cuff will be deflated, but to obtain the final tracings, the participant should lie still for another 5-10 minutes.
Examine whether chronic stress burden and autonomic dysfunction during daily life is elevated in CMD women. | At the end of 1 week of monitoring
  The research team will compare anginal symptoms, chronic and daily life stress, and autonomic function measured during one week of home monitoring between CMD and the two control groups. Participants will use a smartphone to track their symptoms and stress.

OTHER OUTCOMES:
Stressor frequency over 7 days | At the end of 1 week of monitoring
  Participants will use the Actiwatch® Spectrum Pro (Philips-Respironics, Inc.) wristwatch-style actigraphs containing a calibrated accelerometer that records movement activity in discrete epochs and detects physical activity as well as onset and offset of sleep. It provides sleep quality parameters which will be a useful addition to our analysis, as sleep quality is related to stress.
Assessment of quality of life and relationship to anginal symptoms | Baseline and 12 months
  Anginal symptoms and quality of life will be assessed at 12 months of follow-up. MACE and angina hospitalization will also be obtained. Participants will complete the Seattle Angina Questionnaire (SAQ). SAQ asks questions about daily activities and how many limitations they experience due to chest pain, chest tightness, or angina over the past 4weeks. Scored by assigning each response an ordinal value, beginning with 1 for the response that implies the lowest level of functioning, and summing across items within each of the five scales. Scale scores are then transformed into a 0- 100 range by subtracting the lowest possible scale score, dividing by the range of the scale, and multiplying by 100. Because each scale monitors a unique dimension of coronary artery disease, no summary score is generated.
Assessment of general health status | Baseline and 12 months
  SF-36v2 Health Survey measures functional health and well-being from the patient's point of view. It consists of eight scales yielding two summary measures: physical and mental health. The physical health measure includes four scales of physical functioning, role-physical, bodily pain, and general health. The mental health measure is composed of vitality, social functioning, role-emotional, and mental health. A final item, termed self-reported health transition, is answered but is not included in the scoring process. The SF-36 offers a choice of recall format: standard (4 weeks) or acute (1 week) time frame. Likert scales and yes/no options are used to assess function and well-being. To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
Changes in injury and inflammation biomarker with mental stress among the three groups. | Baseline and at the end of the mental stress test
  The research team will administer questionnaires and different types of mental stress tests, including a speech task over a situation that made participant upset or angry, and/or a math test. Blood will be drawn to measure inflammatory biomarker.
Changes in catecholamines (norepinephrine and epinephrine) with mental stress among the three groups. | Baseline and during mental stress test
  The research team will administer questionnaires and different types of mental stress tests, including a speech task over a situation that made you upset or angry, and/or a math test. Blood will be drawn to measure stress hormones.

CONTACTS AND LOCATIONS:
Overall Officials: Puja K Mehta, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory Hospital Midtown, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Emory Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
The research team will share de-identified group demographic data and outcomes with the sponsor and other researchers who request access.
Supporting Information: Study Protocol, SAP
Time Frame: The research team will share the data after the study completion and after the initial data is published.
Access Criteria: The research team will share the data via secure data transfer